CLINICAL TRIAL: NCT03893812
Title: Combined Role of Color Doppler and Diffusion Weighted MRI In Differentiation Between Benign and Malignant Tumors of Major Salivary Glands
Brief Title: Color Doppler and Mri Diffusion in Major Salivary Gland Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Alam El-Din, Principal Investigator, Assiut University
Other Study IDs: doppler & MRdiffusion salivary
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Salivary Gland Diseases
MeSH Terms: conditions — Salivary Gland Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — diffusion weighted MR
Device: Ultrasound — Color Doppler ultrasound

SUMMARY:
This study intend to evaluate the combined value of ADC and COLOR DOPPLER in differentiating benign and malignant salivary gland tumors in comparison to histopathological findings and its use in preoperative prediction of benign and malignant masses.

DETAILED DESCRIPTION:
the study aim to achieve preoperative differentiation between benign and malignant masses of the major salivary glands using the ADC values and Color Doppler values (PSV - PI - RI)

ELIGIBILITY:
Inclusion Criteria:

1- patients must be 18 of age or older. 2= patients must have a suspicious swelling in major salivary glands.

Exclusion Criteria:

1. Patients with history of metal plates or screws or artificial joints.
2. Patients who have phobia of indoor places.
3. Patients with contraindication to MRI like intra-cerebral aneurysmal clips, cardiac pacemaker, and metallic foreign body at region of examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a suspicious swelling in major salivary glands.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The ADC values and Color Doppler values (PSV-PI-RI) of major salivary gland masses | baseline
  The ADC values and Color Doppler values (PSV-PI-RI) of major salivary gland masses will differ according to the nature of the mass determined by histopathological finding